CLINICAL TRIAL: NCT01184781
Title: Prospective Comparison of Capsule Endoscopy Pillcam II™ Versus Colonoscopy for the Detection of Adenomatous Polyps and Cancer in a High Risk Population
Brief Title: Project PREVAM : Prospective Comparison of Capsule Endoscopy Pillcam II™ Versus Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-PP-02
Record Dates: First submitted 2010-07-26; First posted 2010-08-19 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Adenomatous Polyps; Cancer
MeSH Terms: conditions — Adenomatous Polyps; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): On the same patient, we compare both methods (video-colonoscopy vs capsule endoscopy)
  Interventions: Device: Comparison of capsule endoscopy Pillcam II™ versus colonoscopy

INTERVENTIONS:
Device: Comparison of capsule endoscopy Pillcam II™ versus colonoscopy — On the same patient, we compare both methods (video-colonoscopy vs capsule endoscopy)

SUMMARY:
The aim of the study is to perform a prospective, multicenter research comparing capsule endoscopy with the video colonoscopy in the detection of the adenomatous polyps and cancer specifically in a high risk population (sensibility, specificity, NPV, PPV and diagnostic accuracy). The investigators will used the Pillcam II™ colon capsule (second generation) and a high resolution colonoscope (with high definition). Both procedures will be perform in the same day with an adapted bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient with 40 years old and first degree relative affected by colo rectal cancer at age ≥ 60 ans
* Patient with 40 years old or ten years before the age at affected disease in case or first deree relative colo rectal cancer before 60 years old.
* Fecal occult blood test positive
* Personal history of adenomatous polyps
* Personnal history of acromegaly
* Patient with social insurance
* Persons already participating in another clinical trial..
* Signature of informed consent

Exclusion Criteria:

* Pregnancy or breast feeding woman
* Déficience mentale du sujet rendant sa participation à l'essai impossible
* Pacemaker or all electronic devices implanted
* Patient with swallowing disorder, or digestive stricture know or suspected by the investigator
* Previous history of intestinal surgery, radiotherapy or inflammatory bowel disease
* Previous history of polyadenomatous congenital disease, Lynch syndrome
* Intolerance with dompéridon and/or bisacodyl
* Intolerance with oral intake of NaP, polyethylen glycol (PEG) or macrogol
* Colonoscopy contre indication for anesthesiologic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 7 days
  The investigators want to know if the capsule endoscopie is more or less effective than colonoscopy to detect lesion or abdominal cancer.

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 7 days
  Presence of at least one polyp at capsule endoscopy and colonoscopy with both operators unaware of each other's findings until completion of the procedures.
  Comparison of the different class of size for all polyps Comparison of Kudo and Paris classification of the polyps at endoscopy capsule and colonoscopy Tolerance, pain and discomfort between the both procedure Acceptability of both procedure at day 1 and day 7 Accuracy of the localization of the polyp or the lesion at the capsule endosocpy comparated with the colonoscopy topography (Gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: HEBUTERNE Xavier, PU-PH, Study Director — Digestive department
Locations (2):
- Digestive department - Archet hospital, Nice, France
- Gastro entérology department, Sanremo, Italy

REFERENCES:
- [Derived] Parodi A, Vanbiervliet G, Hassan C, Hebuterne X, De Ceglie A, Filiberti RA, Spada C, Conio M. Colon capsule endoscopy to screen for colorectal neoplasia in those with family histories of colorectal cancer. Gastrointest Endosc. 2018 Mar;87(3):695-704. doi: 10.1016/j.gie.2017.05.023. Epub 2017 May 26. PMID 28554656